CLINICAL TRIAL: NCT00792688
Title: Double-Blind, Randomized, Placebo-Controlled Phase 2 Study to Investigate the Safety and Efficacy of 0.1% and 1.0% Topically Applied GLYC-101, Compared to Placebo, in Patients Undergoing Carbon Dioxide Laser Skin Resurfacing of the Lower Eyelids.
Brief Title: Efficacy Study of GLYC-101 to Evaluate Outcomes After Laser Ablation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: TR Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GLYC-101-1b
Record Dates: First submitted 2008-11-14; First posted 2008-11-18 (Estimated); Results first posted 2011-07-25 (Estimated); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Wounds
Keywords: burn wounds; wound healing
MeSH Terms: conditions — Wounds and Injuries; Burns

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- 1 (Experimental): GLYC-101 Gel, 0.1% on one eyelid and Placebo Gel on the other eyelid
  Interventions: Drug: GLYC-101 Gel (0.1%); Drug: GLYC-101 Placebo
- 2 (Experimental): GLYC-101 Gel, 1.0% on one eyelid and Placebo Gel on the other eyelid
  Interventions: Drug: GLYC-101 Gel (1.0%); Drug: GLYC-101 Placebo
- 3 (Experimental): GLYC-101 Gel, 0.1% on one eyelid and GLYC-101 Gel, 1.0% on the other eyelid
  Interventions: Drug: GLYC-101 Gel (0.1%); Drug: GLYC-101 Gel (1.0%)

INTERVENTIONS:
Drug: GLYC-101 Gel (0.1%) — Topical administration to the laser-ablated area on days 1 (day of laser ablation), 2, 3, 4, and 5.
  Arms: 1; 3
Drug: GLYC-101 Gel (1.0%) — Topical administration to the laser-ablated area on days 1 (day of laser ablation), 2, 3, 4, and 5.
  Arms: 2; 3
Drug: GLYC-101 Placebo — Topical administration to the laser-ablated area on days 1 (day of laser ablation), 2, 3, 4, and 5.
  Arms: 1; 2

SUMMARY:
The primary objectives of this study are to evaluate safety and efficacy of topically applied Glucoprime gel (GLYC-101, 0.1% and GLYC-101, 1.0%) in promoting wound healing in cosmetic surgery patients undergoing Carbon Dioxide Laser Skin Resurfacing (CO2 LSR) of the lower eyelids. The study will observe the effects of the topical agent over the course of 1 month following the initial treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male and female healthy volunteer subjects, between 25 and 70 years of age, giving informed consent for facial laser ablation of the lower eyelid areas for the purpose of wrinkle removal.
* Lower eyelid skin is free of any irritation, scarring or dermatologic conditions which might interfere with the study.
* Willing and able to participate in the study and follow all study directions.
* Able to read, understand and sign the consent form prior to any study related procedures.

Exclusion Criteria:

* Female subjects who are pregnant, nursing, or planning a pregnancy during the course of the study, as determined by the interview and a urine pregnancy test.
* Presence of irritation or dermatologic skin conditions in the lower eyelid area.
* Known allergies to materials within the test formulations (i.e., yeast and/or yeast products).
* Use of topical or systemic drugs (corticosteroids, retinoids, immune modulators, immune suppressants, drugs with potential for contact dermatitis, drugs with potential for skin discoloration) that may have an effect on wound healing or may impact skin pigmentation.
* A history, upon wounding, of developing thickened scars, keloids, or excessive pigment change.
* An unstable or severe inter-current medical condition that, in the opinion of the investigator, might interfere with interpretation of study results or render the subject at high risk for treatment complications.
* Use of any investigational medication or device for any indication within 30 days of screening.

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2008-10; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Joseph, MD, Principal Investigator — The Clinical Testing Center of Beverly Hills
Locations (1):
- CLINICAL TESTING CENTER of BEVERLY HILLS, Beverly Hills, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment started in October 2008 and ended in 2009 at a single site, Clinical Testing Center of Beverly Hills, Beverly Hills, California, United States, 90210.
Pre-assignment Details: All subjects needed to meet specific inclusion and exclusion criteria as described in the Eligibility Criteria section. Eligible subjects were randomly assigned to receive GLYC-101 0.1%, GLYC-101 1%, or placebo.
Groups:
- GLYC-101 Gel, 0.1% on One Eyelid & Placebo on the Other Eyelid: GLYC-101 Gel (0.1%) Topical administration to the laser-ablated area on Days 1 (day of laser ablation), 2, 3, 4, and 5.
  Placebo Gel Topical administration to the laser-ablated area on Days 1 (day of laser ablation), 2, 3, 4, and 5.
- GLYC-101 Gel, 1.0% on One Eyelid & Placebo on the Other Eyelid: GLYC-101 Gel (1%) Topical administration to the laser-ablated area on Days 1 (day of laser ablation), 2, 3, 4, and 5.
  Placebo Gel Topical administration to the laser-ablated area on Days 1 (day of laser ablation), 2, 3, 4, and 5.
- GLYC-101 Gel 0.1% on 1 Eyelid & GLYC-101 Gel 1.0% on the Other: GLYC-101 Gel (0.1%) Topical administration to the laser-ablated area on Days 1 (day of laser ablation), 2, 3, 4, and 5.
  GLYC-101 Gel (1%) Topical administration to the laser-ablated area on Days 1 (day of laser ablation), 2, 3, 4, and 5.
Period: Overall Study
Arm/Group | GLYC-101 Gel, 0.1% on One Eyelid & Placebo on the Other Eyelid | GLYC-101 Gel, 1.0% on One Eyelid & Placebo on the Other Eyelid | GLYC-101 Gel 0.1% on 1 Eyelid & GLYC-101 Gel 1.0% on the Other
Started | 9 | 8 | 9
Completed | 9 | 8 | 9
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GLYC-101 Gel, 0.1% on One Eyelid & Placebo on the Other Eyelid | GLYC-101 Gel, 1.0% on One Eyelid & Placebo on the Other Eyelid | GLYC-101 Gel 0.1% on 1 Eyelid & GLYC-101 Gel 1.0% on the Other | Total
Number analyzed (Participants) | 9 | 8 | 9 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 9 | 7 | 8 | 24
  >=65 years | 0 | 1 | 1 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.1 (7.98) | 46.4 (12.83) | 53.3 (9.41) | 51.1 (10.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 6 | 22
  Male | 1 | 0 | 3 | 4
Region of Enrollment [Number; unit: participants]
  United States | 9 | 8 | 9 | 26

OUTCOME MEASURES:

1. Primary Outcome: Time to Complete Wound Closure (Epithelialization)
Description: Subjects were evaluated daily from the time of the laser procedure and initial application of test article until the subject's wounds reached 100% epithelialization. Efficacy was assessed based on the time to complete epithelialization in terms of the number of days from Day 1 (day of laser ablation) to the day on which complete epithelialization was observed.
Time Frame: Over the course of 1 month following the initial treatment.
Population: Analysis was Per Protocol.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | All Treatments GLYC-101 Gel, 0.1% | All Treatments GLYC-101 Gel, 1.0% | All Treatments Placebo
Number analyzed (Participants) | 18 | 17 | 17
days | 10.9 (5.17) | 13.1 (8.31) | 16.3 (9.93)
Statistical Analysis 1: Comparison: All Treatments GLYC-101 Gel, 0.1% vs All Treatments Placebo; Test type: Superiority or Other; p = 0.0062, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: All Treatments GLYC-101 Gel, 1.0% vs All Treatments Placebo; Test type: Superiority or Other; p = 0.0331, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Cosmesis/11-point Likert Scale
Description: The cosmetic effect on each lower eyelid using an 11-point Likert Scale (0 = not healed and 10 = healed).
Time Frame: At 1 month following the initial treatment.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | All Treatments GLYC-101 Gel, 0.1% | All Treatments GLYC-101 Gel, 1.0% | All Treatments Placebo
Number analyzed (Participants) | 18 | 17 | 17
scores on a scale | 8.9 (1.28) | 8.6 (1.17) | 8.5 (1.50)

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected over the course of 1 month.
Description: AEs were collected at baseline and each study visit.
Arm/Group | GLYC-101 Gel, 0.1% on One Eyelid & Placebo on the Other Eyelid | GLYC-101 Gel, 1.0% on One Eyelid & Placebo on the Other Eyelid | GLYC-101 Gel 0.1% on 1 Eyelid & GLYC-101 Gel 1.0% on the Other
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/8 | 1/9
Other Adverse Events (participants affected / at risk) | 9/9 | 8/8 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GLYC-101 Gel, 0.1% on One Eyelid & Placebo on the Other Eyelid (N=9) | GLYC-101 Gel, 1.0% on One Eyelid & Placebo on the Other Eyelid (N=8) | GLYC-101 Gel 0.1% on 1 Eyelid & GLYC-101 Gel 1.0% on the Other (N=9)
HIV test positive (Investigations) | 0 (0) | 0 (0) | 1 (1) — This Serious Adverse Event is not related to study drugs.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GLYC-101 Gel, 0.1% on One Eyelid & Placebo on the Other Eyelid (N=9) | GLYC-101 Gel, 1.0% on One Eyelid & Placebo on the Other Eyelid (N=8) | GLYC-101 Gel 0.1% on 1 Eyelid & GLYC-101 Gel 1.0% on the Other (N=9)
Application site pain (General disorders) | 9 (70) | 8 (62) | 9 (71)
Impaired healing (General disorders) | 2 (4) | 1 (1) | 1 (2)
Procedural pain (Injury, poisoning and procedural complications) | 6 (11) | 5 (14) | 6 (13)
Chemical eye injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Eye pruritus (Eye disorders) | 4 (11) | 3 (7) | 6 (10)
Conjunctivitis (Eye disorders) | 0 (0) | 1 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period of up to 90 days. The sponsor can require changes to the communication to remove any confidential information.